CLINICAL TRIAL: NCT06455423
Title: Supplemental Effects of ELDOA in Addition to Thoracic Manipulation on Upper Back Pain, Thoracic Kyphosis and Forward Head Posture in Thoracic Hypomobility (The ELDOA-MAN Study)
Brief Title: Supplemental Effects of ELDOA in Addition to Thoracic Manipulation on Upper Back Pain, Thoracic Kyphosis and Forward Head Posture in Thoracic Hypomobility
Acronym: ELDOA-MAN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/15
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Forward Head Posture; Thoracic Hypomobility; Upper Back Pain
MeSH Terms: conditions — Back Pain | interventions — Exercise; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The study will consist of two groups.
Who Masked: Investigator
Masking Description: The investigator will be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAN group (Active Comparator): the standard MAN group will only receive thoracic manipulation and physical therapy
  Interventions: Procedure: Thoracic Manipulation; Procedure: Chin tuck in exercises; Procedure: Thoracic Extension Exercise; Procedure: Scapular Retraction Exercises; Device: Hot Pack; Device: TENS
- ELDOA-MAN group (Experimental): The ELDOA-MAN group will receive ELDOA exercises in addition to thoracic manipulation and physical therapy.
  Interventions: Procedure: Thoracic Manipulation; Procedure: Chin tuck in exercises; Procedure: Thoracic Extension Exercise; Procedure: Scapular Retraction Exercises; Device: Hot Pack; Device: TENS; Procedure: ELDOA

INTERVENTIONS:
Procedure: Thoracic Manipulation — Thoracic manipulation will be administered at hypomobile or stiff segments.
Procedure: Chin tuck in exercises — Chin tuck in exercises
Procedure: Thoracic Extension Exercise — Thoracic Extension Exercise
Procedure: Scapular Retraction Exercises — Scapular Retraction Exercises
Device: Hot Pack — Hot Pack
Device: TENS — Trans Cutaneous Electric Nerve Stimulation (TENS)
Procedure: ELDOA — ELDOA exercises
  Arms: ELDOA-MAN group

SUMMARY:
The purpose of this study is to determine the supplemental effects of ELDOA in addition to thoracic manipulation on upper back pain, thoracic kyphosis and forward head posture in thoracic hypomobility.

ELIGIBILITY:
Inclusion Criteria:

* Both male and females
* Adults (19-44 years)
* Upper back pain or discomfort
* Forward head posture
* Thoracic hypomobility
* Thoracic hyperkyphosis

Exclusion Criteria:

* Ankylosing spondylitis
* History of Spinal Fusion or spinal surgery (discectomy/laminectomy etc.)
* Degenerative disc disorders, Facet joint syndrome
* Cervical radiculopathy, Scoliosis
* Spinal Stenosis or Myelopathy
* Recent fracture or surgery
* TB of spine, Spondylolisthesis
* Not able to attend regular therapy appointments
* Fibromyalgia/myofascial pain syndrome

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Upper Back Pain or Discomfort | 3 weeks
  Upper Back Pain or Discomfort will be quantified using Visual Analogue Scale. A higher score signifies greater pain or discomfort on a 0-100mm line.
Thoracic Kyphosis | 3 weeks
  Thoracic Kyphosis will be quantified using an inclinometer. A higher score signifies increased Kyphosis.
Thoracic Range of Motion (ROM) | 3 weeks
  Thoracic Range of Motion (ROM) will be quantified using an inclinometer. A higher score signifies greater mobility of thoracic spine.
Forward Head Posture | 3 weeks
  Forward Head Posture will be quantified via Craniovertebral Angle (CVA). A smaller CVA indicates increased forward head posture.
Functional ability | 3 weeks
  Functional ability will be quantified using Spine Functional Index (SFA). A smaller SFA score indicates greater functional ability.

CONTACTS AND LOCATIONS:
Overall Officials: Samra Batool, Principal Investigator — Foundation University Islamabad; Muhammad Osama, Study Chair — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No